CLINICAL TRIAL: NCT02009267
Title: Nuss Procedure: Clinical Options in Pediatric Pain Management?
Status: Completed | Type: Observational
Sponsor: Ralph Beltran (Other)
Responsible Party: Sponsor-Investigator, Ralph Beltran, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00702
Record Dates: First submitted 2013-11-19; First posted 2013-12-11 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient controlled analgesia: Use of patient controlled analgesia (PCA) for the management of postoperative pain after the Nuss procedure.
  Interventions: Device: Patient controlled analgesia
- Continuous thoracic epidural infusion: Continuous thoracic epidural infusions (TE) for the management of postoperative pain after the Nuss procedure.
  Interventions: Procedure: Continuous thoracic epidural infusions
- Continuous paravertebral blockade: Continuous paravertebral blockade (PVB) for the management of postoperative pain after the Nuss procedure.
  Interventions: Procedure: Continuous paravertebral blockade

INTERVENTIONS:
Device: Patient controlled analgesia — A programable electronically controlled infusion pump that delivers an amount of intravenous analgesic when the patient presses a button.
  Groups: Patient controlled analgesia
Procedure: Continuous thoracic epidural infusions — Continuous thoracic epidural infusions (TE) involves continuous infusion of drugs through a catheter placed into the epidural space, resulting in a loss of sensation-including the sensation of pain-by blocking the transmission of signals through nerve fibers in or near the spinal cord.
  Groups: Continuous thoracic epidural infusion
Procedure: Continuous paravertebral blockade — Continuous paravertebral blockade (PVB) is the technique of injecting local anesthetic adjacent to the thoracic vertebra that anesthetizes the spinal nerve roots after they exit the spinal canal.
  Groups: Continuous paravertebral blockade

SUMMARY:
A retrospective chart review study analyzing the benefits of patient controlled analgesia, thoracic epidural analgesia, and paravertebral nerve block catheters in patients having surgical repair of pectus excavatum using the Nuss procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing the NUSS procedure since the beginning of 2011 to Sept. 30th, 2013.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing the Nuss procedure to correct pectus excavatum at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total morphine dose | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Total morphine dose will be evaluated in mg/kg/24 hour period, beginning with post-op day 0 until discharge from the hospital.

SECONDARY OUTCOMES:
Pain score | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Pain scores obtained from the visual analog scale.
Length of hospitalization | Within the first week after surgery.
  Determine if there is a difference in length of hospitalization, and time to discharge.
Nausea and vomiting | 0-48 hrs. post-op
  Determine the incidence of nausea and vomiting measured by the postoperative ondansetron dosing, beginning with arrival to floor and up to the first 48 hrs of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Beltran Ralph, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States